CLINICAL TRIAL: NCT05491200
Title: COMPARE STEMI ONE- Comparison Of Reduced DAPT Followed by P2Y12 Inhibitor Monotherapy With Prasugrel vs stAndard Regimen in STEMI Patients Treated With OCT-guided vs aNgio-guided completE Revascularization
Brief Title: Comparison Of Reduced DAPT Followed by P2Y12 Inhibitor Monotherapy With Prasugrel vs stAndard Regimen in STEMI Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Research Maatschap Cardiologen Rotterdam Zuid (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RM21
Record Dates: First submitted 2022-08-02; First posted 2022-08-08 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: ST Elevated Myocardial Infarction; Dual Antiplatelet Therapy
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Prasugrel-based short DAPT (Experimental): Prasugrel-based short DAPT (30-45 days) followed by Prasugrel monotherapy for 11 months.
  Interventions: Drug: Prasugrel based short DAPT
- Prasugrel based standard DAPT (Active Comparator): Prasugrel-based DAPT for 1 year
  Interventions: Drug: Prasugrel based standard DAPT
- OCT guided non-culprit lesion (Experimental): Complete revascularization of non culprit lesions guided by OCT
  Interventions: Device: OCT guided revascularization
- Angio guided non-culprit lesion (Active Comparator): Complete revascularization of non culprit lesions guided by Angio
  Interventions: Device: Angio guided revascularization

INTERVENTIONS:
Drug: Prasugrel based short DAPT — Prasugrel-based short DAPT (30-45 days) followed by Prasugrel monotherapy versus
  Arms: Prasugrel-based short DAPT
Drug: Prasugrel based standard DAPT — Prasugrel based DAPT for 1 year
  Arms: Prasugrel based standard DAPT
Device: OCT guided revascularization — OCT guided revascularization of the non-culprit lesions
  Arms: OCT guided non-culprit lesion
Device: Angio guided revascularization — Angio guided revascularization of the non-culprit lesions
  Arms: Angio guided non-culprit lesion

SUMMARY:
The study is a multi-centre, Open-label, Randomized Controlled, 1:1 trial comparing Prasugrel-based short DAPT (30-45 days) followed by Prasugrel monotherapy versus standard DAPT regimen in STEMI patients in terms of safety and efficacy endpoints.

In the subgroup of STEMI patients with MVD, a sub-randomization will allow a comparison between a complete revascularization OCT-guided versus complete revascularization angiography-guided stent in terms of efficacy and safety endpoints.

DETAILED DESCRIPTION:
Consecutive patients with STEMI planned for pPCI will be screened for eligibility criteria and treated as per standard of care with ASA and Prasugrel 60 mg loading dose. The culprit lesion will be treated during the index procedure. Non culprit lesions in patients with MVD will be treated during staged procedure(s), in any case last instalment of staged procedure(s) should be scheduled within 15 days after index procedure. Complete revascularization of non culprit lesions will be allocated to either OCT- or angio-guided strategy (OCT randomization). At 30-45 days follow-up after index procedure, if inclusion criteria are met, patients will be randomized to prasugrel monotherapy or standard DAPT regimen (DAPT randomization).

The follow-up duration is 35 months after DAPT randomization, i.e. clinical outcomes will be analysed at 11 and 35 months after DAPT randomization.

ELIGIBILITY:
Inclusion Criteria:

Eligibility at index procedure

All STEMI patients who are planned to be treated with PCI:

ST segment elevation myocardial infarction

Chest discomfort suggestive of cardiac ischemia ≥20 min at rest with 1 of the following ECG features:

* ST segment elevation ≥2 contiguous ECG leads
* new or presumably new left bundle branch block

In patients with multivessel disease, treatment only of the culprit lesion / target vessel during primary PCI is recommended.

Eligibility at 30-45 days

* All patients who have provided informed consent
* Compliance to DAPT with no regimen modifications (Non-adherence Academic Research Consortium 0)
* No occurrence of significant event (such as MI, unplanned revascularisation, stent thrombosis, stroke, major vascular complication/bleeding BARC Types 3 or greater).
* Successful revascularization: - Successful delivery and deployment of the Study device(s), with final residual stenosis of <30% (visually) for all target lesions.
* Complete revascularization performed when more than 1 significant lesion, during the index procedure or in staged procedure(s) occurring within 15 days from the index procedure. Physiologic assessment highly recommended for lesions with stenosis between 50% and 90%.

Exclusion criteria

* Patients on oral anticoagulation
* Contraindication to P2Y12 inhibitors and/or to Cardioaspirin or to any of the excipients (hypersensitivity, history of any stroke or transient ischemic attack within the last 12 months, active bleeding or haemorrhagic diathesis, fibrin-specific fibrinolytic therapy less than 24 h before randomization, severe hepatic dysfunction (Child-Pugh C), history of asthma induced by the administration of salicylates or substances with a similar action, notably non-steroidal anti-inflammatory medicines, history of gastrointestinal perforation or acute gastrointestinal ulcers, severe cardiac failure (NYHA grade III or IV), combination with methotrexate at doses of 15 mg/week or more).
* Patients who have received P2Y12 inhibitors other than Prasugrel in the ambulance (Ticagrelor or Clopidogrel loading dose) or are already on P2Y12 inhibitors, may be enrolled in the protocol, provided that the Prasugrel loading dose is administered at admission, according to current guidelines recommendations (see section 5.2.2).
* Concomitant oral or i.v. therapy with strong CYP3A inhibitors (e.g., ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir, grapefruit juice >1L/day), CYP3A substrates with narrow therapeutic indices (e.g., cyclosporine, quinidine), or strong CYP3A inducers (e.g., rifampin), - rifampicin, phenytoin, carbamazepine, dexamethason, phenobarbital
* Platelet count <100.000/μL at the time of screening
* Anemia (hemoglobin <10 g/dL) at the time of screening
* Comorbidities associated with life expectancy <1 year
* Pregnancy, giving birth within the last 90 days, or lactation (see appendix III for women of childbearing potential)
* PCI indication for stent thrombosis or previous history of definite stent thrombosis
* Non-deferrable major surgery on DAPT after PCI
* Cardiogenic shock
* Out of hospital cardiac arrest (OHCA) unless survivors of ventricular arrythmia with prompt return of spontaneous circulation (ROSC)
* Patients with severe renal impairment: creatinine clearance ≤30 ml/min/1.73 m2 (as calculated by MDRD formula for estimated GFR).
* Patients participating in another interventional (device of drug trial) within the previous 12 months or patients to whom an investigational drug was administered in the 30 days prior to screening, or 5 half-lives of the study drug, whichever is longer.
* No informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1656 (Estimated)
Dates: Start 2022-07-22 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
non inferiority of a Prasugrel-based short DAPT (30-45 days) followed by Prasugrel 11 month monotherapy versus standard 12 month DAPT regimen | 11 months
  Incidence of Net Adverse Clinical Events (NACE) at 11 months post DAPT randomization as composite of all cause death, MI, stroke or BARC bleeding 3 or 5
superiority of an Optical Coherence Tomography (OCT)-guided revascularization completion as compared to a standard angiography-guided revascularization completion. | immediately after the procedure
  Post-procedural Minimal Stent Area (MSA)

SECONDARY OUTCOMES:
Composite of MACCE | 3 year
  Composite of the number of major adverse cardiac and cerebrovascular events (MACCE) defined as cardiovascular death, myocardial infarction, or ischaemic stroke
BARC type 3 or 5 events | 1 and 3 years
  Number of BARC type 3 or 5 events occuring

CONTACTS AND LOCATIONS:
Overall Officials: Valeria Paradies, MD, PhD, Principal Investigator — Research Maatschap Cardiologen Rotterdam Zuid
Locations (26):
- Belgium (5):
  - Imelda Bonheiden, Bonheiden
  - AZ St.Jan, Bruges
  - ZOL Genk, Genk
  - UZ Leuven, Leuven
  - AZ Delta, Roeselare
- Czechia (3):
  - FN BRNO, Brno
  - Masaryk Hospital Usti nad Labem -, Hradec Králové
  - Charles University Hospital, Prague
- Germany (3):
  - Asklepios Klinik Bad Oldesloe, Bad Oldesloe
  - Segeberger Kliniken, Bad Segeberg
  - University hospital Dresden, Dresden
- Italy (6):
  - Ospedale Papa Giovanni XXIII, Bergamo
  - University of Ferrara, Ferrara
  - University San Martino, Genova
  - Centro Cardiologico Monzino IRCCS, Milan
  - University Federico II, Napoli
  - University Gemelli, Roma
- Netherlands (6):
  - Albert Schweitzer ziekenhuis, Dordrecht
  - Catherina ziekenhuis, Eindhoven
  - RadboudUMC, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - Maasstadziekenhuis, Rotterdam
  - Haga hospital, The Hague
- Serbia (3):
  - Institute for CVD Dedinje, Belgrade
  - University clinical center of Serbia, Belgrade
  - Institute for CVD Vojvodine, Kamenitz

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paradies V, Van Mieghem NM, Oemrawsingh RM, Richardt G, Esposito G, Campo G, Burzotta F, Canova P, Linke A, Porto I, Trabattoni D, Teeuwen K, Adriaenssens T, Kala P, Stankovic G, Vliet RV, Giacoppo D, Daemen J, Smits PC. Prasugrel monotherapy versus standard DAPT in STEMI patients with OCT-guided or angio-guided complete revascularisation: design and rationale of the randomised, multifactorial COMPARE STEMI ONE trial. EuroIntervention. 2025 May 16;21(10):571-580. doi: 10.4244/EIJ-D-24-00829. PMID 40375771